CLINICAL TRIAL: NCT01340105
Title: Microwave Versus Radiofrequency Ablation for Hepatocellular Carcinoma: a Prospective Randomized Control Trial
Brief Title: Effectiveness of Microwave Ablation of Hepatocellular Carcinoma as Compared to Radiofrequency Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cheung Yue Sun, Associate Consultant, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT11005
Record Dates: First submitted 2011-04-19; First posted 2011-04-22 (Estimated); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Microwave ablation; Radiofrequency ablation; Randomised controlled trial
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiofrequency Ablation

ARMS (2):
- Microwave (Experimental): Hepatocellular carcinoma treated with microwave ablation
  Interventions: Procedure: Microwave ablation
- Radiofrequency (Active Comparator): Hepatocellular carcinoma treated with radiofrequency ablation
  Interventions: Procedure: Radiofrequency ablation

INTERVENTIONS:
Procedure: Microwave ablation — Use of microwave energy to ablate hepatocellular carcinoma. It can be employed by percutaneous, open surgery or laparoscopic means.
  Arms: Microwave
Procedure: Radiofrequency ablation — Use of radiofrequency energy to ablate hepatocellular carcinoma. It can be employed by percutaneous, open surgery or laparoscopic means.
  Arms: Radiofrequency

SUMMARY:
The purpose of this study is to compare microwave ablation using the Acculis Microwave Tissue Ablation (MTA) System with conventional radiofrequency ablation (RFA) using Covidien cool-tip radiofrequency needle in patients with localized unresectabe hepatocelluar carcinoma (HCC).

The investigators hypothesize that microwave ablation can achieve a better complete ablation rate as compared to radiofrerquency ablation.

A randomized comparative study is performed by randomly assigned participants to microwave ablation arm or radiofrequency ablation arm. The efficacy of treatment outcome is assessed by the complete tumor ablation rate at 1 month, recurrence rate and survival time of participants. Safety of the procedures is also compared between the 2 treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Unresectable hepatocellular carcinoma (HCC) and tumor amendable for local ablation
* Resectable HCC but patient opts for local ablation
* Maximum diameter of tumor ≤6cm
* Maximum number of tumor nodules ≤3
* Absence of radiology evidence of major vascular or bile duct invasion
* Child's A or B liver function
* Karnofsky performance status ≥70%

Exclusion Criteria:

* Informed consent not available
* Pregnant female patients
* Tumors unfavourable for local ablation (e.g. tumor close to porta hepatis)
* HCC with history of rupture
* Concomitant hepatectomy
* Patients with chronic renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Complete ablation rate | 1 month
  Measure by post-ablation Computed Tomography (CT) with reference to alpha-fetoprotein (AFP)

SECONDARY OUTCOMES:
Treatment related mortality | 30-day
  Mortality within 30 days after operation
Recurrent disease | 3 year
  It is defined as the imaging detected new lesions
Survival | 3 year
  Overall and disease-free survival
Long-term liver function | 3 year
  Monitoring of liver function test result and the occurrance of decompensated cirrhosis
Treatment related morbidity | 30-day
  Complications related to the treatment received
Hospital stay | 30-day
  Total length of hospital stay (days)

CONTACTS AND LOCATIONS:
Overall Officials: Kit-fai Lee, MBBS, Principal Investigator — Department of Surgery, The Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No